CLINICAL TRIAL: NCT05940194
Title: A Phase 1/2 Randomized, Active- Controlled, Observer-blind Trial to Assess the Safety and Immunogenicity of COVIVAC Vaccine Produced by IVAC in Adults ≥ 18 and ≥ 60 Years Old in Vietnam
Brief Title: NDV-HXP-S Vaccine Clinical Trial (COVIVAC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Vaccines and Medical Biologicals, Vietnam (Industry)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other); Center for Disease Control of Thai Binh Province, Vietnam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: COVIVAC-0102 (Phase 2)
Record Dates: First submitted 2023-07-08; First posted 2023-07-11 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- COVIVAC 3 mcg (Experimental): 3 mcg IVAC COVIVAC vaccine for intramuscular injection administered as two doses (0.5mL each) 28 days apart.
  Interventions: Biological: COVIVAC vaccine
- COVIVAC 6 mcg (Experimental): 6 mcg IVAC COVIVAC vaccine for intramuscular injection administered as two doses (0.5mL each) 28 days apart.
  Interventions: Biological: COVIVAC vaccine
- AZD1222 (Active Comparator): AZD1222 (AstraZeneca) vaccine for intramuscular injection administered as two doses (0.5mL each) 28 days apart.
  Interventions: Biological: COVIVAC vaccine

INTERVENTIONS:
Biological: COVIVAC vaccine — For prevention Covid-19

SUMMARY:
This prospective, single-center, randomized, placebo-controlled (phase 1) and active-controlled (phase 2), observer-blind Phase 1/2 study includes two separate parts.

After completing the phase 1 interim analysis, 2 doses (3mcg and 6mcg) were selected for phase 2.

In Part 2 of this combined Phase 1/2 study, 374 adults aged 18-75 years will be randomized (1:1:1) to AZD1222, or COVIVAC 3 µg being evaluated in Phase 1 or the intermediate dose of COVIVAC 6 µg being selected after consideration of phase 1 results.

DETAILED DESCRIPTION:
In Part 2 of this combined Phase 1/2 study, 374 adults aged 18-75 years will be randomized (1:1:1) to placebo, or COVIVAC 3 µg being evaluated in Phase 1 or the intermediate dose of COVIVAC 6 µg being selected after consideration of phase 1 results. At least one-third of the subjects in Phase 2 will be aged ≥60 years to ensure that adequate safety and immune data will be available from older and elderly adults to inform the selection of the COVIVAC formulation to advance to Phase 3 studies. The Phase 2 cohort will follow the same visit schedule, and undergo the same procedures and assessments, as in Phase 1. In addition, as exploratory objectives, the anti-NDV HN IgG response will be assessed at V1, V3, V5, and V7 in all subjects, and 36 subjects (equally distributed between the two age strata) will be randomly selected in a 1:1:1 ratio to provide additional blood at V1, V5 and V7 to be used to isolate peripheral blood mononuclear cells (PBMCs) for assessment of T-cell-mediated immunity (CMI).

An interim analysis of Phase 2 data will be conducted after the last subject of the Phase 2 cohort completes V6 (D57) as the basis for selecting the optimal formulation of COVIVAC to advance to Phase 3 studies. As was the case for the Phase 1 interim analysis at the same timepoint, the data generated will include unblinded post-dose 1 and dose 2 safety results for review by the DSMB, and immunogenicity results aggregated by treatment group for review by the Sponsor. The DSMB will consider all accumulated safety data from both phases of the study prior to making any recommendation to the Sponsor that it not advance a formulation based on safety concerns. The Sponsor will ultimately select the formulation to advance to Phase 3 that, in addition to having been judged by the DSMB to have an adequate safety and tolerability profile, is optimal based on relative functional immunogenicity and other programmatic considerations such as those noted above.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years old inclusive at the time of randomization.
2. Having no clinically significant acute medical condition, and no chronic medical condition that has not been controlled within 90 days of randomization, as determined by medical history, physical examination, screening laboratory test results, and clinical assessment of the investigator.
3. Has provided written informed consent prior to performance of any study-specific procedure.
4. Has a body mass index (BMI) of 17 to 40 kg/m2, inclusive, at screening.
5. Resides in study site area and is able and willing to adhere to all protocol visits and procedures.
6. If a woman is of childbearing potential age, must not be breastfeeding or be pregnant (based on a negative urine pregnancy test at screening and during the 24 hours prior to receipt of the first dose of IP), must plan to avoid pregnancy for at least 28 days after the last dose of IP, and be willing to use an adequate method of contraception consistently and have a repeated pregnancy test prior to the second (last) dose of IP.

Exclusion Criteria:

1. Use of any investigational medicinal product within 90 days prior to randomization or planned use of such a product during the period of study participation.
2. History of administration of any non-study vaccine within 28 days prior to administration of study vaccine or planned vaccination within 3 months after enrolment.

   Note: receipt of any COVID-19 vaccine that is licensed or granted Emergency Use Authorization in Vietnam during the course of study participation is not exclusionary if administered after Visit 5.
3. Previous receipt of investigational vaccine for SARS or MERS, or any investigational or licensed vaccine that may have an impact on interpretation of the trial results
4. History of hypersensitivity reaction to any prior vaccination or known hypersensitivity to any component of the study vaccine
5. History of egg or chicken allergy
6. History of angioedema
7. History of anaphylaxis (≥ grade 2)
8. Acute illness (moderate or severe) and/or fever (body temperature measured orally ≥38°C)
9. Any abnormal vital sign deemed clinically relevant by the PI
10. Abnormality in screening laboratory test deemed exclusionary by the PI in consultation with the Sponsor
11. A positive serologic test for hepatitis B (HBsAg) or hepatitis C (HCV Ab) (phase 1 only)
12. History of confirmed HIV
13. History of laboratory-confirmed COVID-19
14. History of malignancy, excluding non-melanoma skin and cervical carcinoma in situ
15. Any confirmed or suspected immunosuppressive or immunodeficient state
16. Administration of immunoglobulin or any blood product within 90 days prior to first study injection or planned administration during the study period.
17. Administration of any long-acting immune-modifying drugs (e.g., infliximab or rituximab) or the chronic administration (defined as more than 14 days) of immunosuppressants within six months prior to first study injection, or planned administration during the study period (includes systemic corticosteroids at doses equivalent to ≥ 0.5 mg/kg/day of prednisone; the use of topical steroids including inhaled and intranasal steroids is permitted).
18. History of known disturbance of coagulation or blood disorder that could cause anemia or excess bleeding. (e.g, thalassemia, coagulation factor deficiencies).
19. Recent history (within the past year) or signs of alcohol or substance abuse.
20. Any medical, psychiatric or behavior condition that in the opinion of the PI may interfere with the study objectives, pose a risk to the subject, or prevent the subject from completing the study follow-up.
21. Employee of any person employed by the Sponsor, the contract research organization (CRO), the PI, study site personnel, or site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2021-08-11 (Actual); Primary Completion 2021-10-18 (Actual); Study Completion 2022-03-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- District Health Center of Vu Thu District, Thái Bình, Thai Binh, Vietnam

REFERENCES:
- [Derived] Thiem VD, Anh DD, Ha VH, Van Thom N, Thang TC, Mateus J, Carreno JM, Raghunandan R, Huong NM, Mercer LD, Flores J, Escarrega EA, Raskin A, Thai DH, Van Be L, Sette A, Innis BL, Krammer F, Weiskopf D. Safety and immunogenicity of an inactivated recombinant Newcastle disease virus vaccine expressing SARS-CoV-2 spike: A randomised, comparator-controlled, phase 2 trial. Vaccine. 2025 Jan 12;44:126542. doi: 10.1016/j.vaccine.2024.126542. Epub 2024 Nov 29. PMID 39615342

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The screening and enrollment were conducted from 11 Aug 2021 to 23 August 2021 at the District Health Center of Vu Thu district, Thai Binh province. Total 737 subjects were screened, and 374 subjects were randomized to 3 treatment arms (124 subjects in COVIVAC 3µg arm, 125 subjects in COVIVAC 6µg arm and 125 in the AZD122 arm).
Pre-assignment Details: This is the phase 2 (part 2) of the phase 1/2 trial of COVIVAC vaccine. After providing informed consent, participants were screened and then randomized to receive either of 2 COVIVAC dose or AZD1222 in the 1:1:1 ratio. Each participant received 2 injections with 28 days apart.
Period: Overall Study
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
Started | 124 | 125 | 125
Completed | 122 | 122 | 121
Not Completed | 2 | 3 | 4
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Migrated/Moved from the study area | 2 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222 | Total
Number analyzed (Participants) | 124 | 125 | 125 | 374
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.9 (14.82) | 48.9 (14.27) | 49.8 (14.17) | 49.2 (14.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 58 | 71 | 189
  Male | 64 | 67 | 54 | 185
Race/Ethnicity, Customized [Number; unit: Participants]
  Kinh | 124 | 124 | 125 | 373
  Other | 0 | 1 | 0 | 1
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.29 (2.67) | 22.27 (2.52) | 22.24 (2.55) | 22.27 (2.57)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local and Systemic Solicited AEs by Severity During the First 7 Days After Each Vaccination.
Description: * Local solicited AEs: Pain or tenderness, Swelling or induration, Erythema
  * Systemic solicited AEs: Fever (defined as oral temperature ≥ 38°C), Headache, Fatigue or malaise, Myalgia, Arthralgia, Nausea or vomiting
  * Severity grading: Mild = Causes no or minimal interference with normal daily activities; intervention not indicated; Moderate =Interferes with but does not prevent normal daily activities; intervention indicated; Severe = Prevents normal daily activities; intervention or hospitalization indicated.
Time Frame: 7 days after each vaccination
Population: All participants received at least one vaccination.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
Number analyzed (Participants) | 124 | 125 | 125
percent of participants
  Any solicited AE after any dose | 78.2 [69.9 to 85.1] | 80.0 [71.9 to 86.6] | 88.0 [81.0 to 93.1]
  Mild solicited AE | 77.4 [69.0 to 84.4] | 78.4 [70.2 to 85.3] | 87.2 [80.0 to 92.5]
  Moderate solicited AE | 24.2 [17.0 to 32.7] | 28.0 [20.3 to 36.7] | 46.4 [37.4 to 55.5]
  Severe solicited AE | 1.6 [0.2 to 5.7] | 1.6 [0.2 to 5.7] | 7.2 [3.3 to 13.2]

2. Primary Outcome: Percentage of Participants With Unsolicited AEs by Severity and Relatedness During the First 28 Days After Each Vaccination
Description: * An unsolicited adverse event is any AE reported spontaneously by the subject, observed by the study staff during study visits or those identified during review of medical records or source documents. Solicited AEs with an onset after the seven-day solicitation period will be considered unsolicited AEs
  * Severity grading: Mild = Causes no or minimal interference with normal daily activities; intervention not indicated; Moderate =Interferes with but does not prevent normal daily activities; intervention indicated; Severe = Prevents normal daily activities; intervention or hospitalization indicated.
Time Frame: 28 days after each vaccination
Population: All participants received at least one vaccination.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
Number analyzed (Participants) | 124 | 125 | 125
percent of participants
  Total unsolicited AE after any dose | 29.0 [21.2 to 37.9] | 23.2 [16.1 to 31.6] | 31.2 [23.2 to 40.1]
  Mild unsolicited AE | 10.5 [5.7 to 17.3] | 7.2 [3.3 to 13.2] | 8.8 [4.5 to 15.2]
  Moderate unsolicited AE | 16.9 [10.8 to 24.7] | 18.4 [12.0 to 26.3] | 23.2 [16.1 to 31.6]
  Severe unsolicited AE | 3.2 [0.9 to 8.1] | 0.8 [0.0 to 4.4] | 0.8 [0.0 to 4.4]
  Related unsolicited AE | 0.0 [0.0 to 2.9] | 0.0 [0.0 to 2.9] | 0.0 [0.0 to 2.9]

3. Primary Outcome: Percentage of Participants With SAEs Severity and Relatedness Throughout the Entire Study Period
Description: A SAE is a specific AE that:
  * Results in death.
  * Is life-threatening.*
  * Requires inpatient hospitalization or prolongation of an existing hospitalization.**
  * Results in a persistent or significant disability or incapacity.***
  * Results in a congenital anomaly or birth defect.
Time Frame: From the first vaccination until Day 197
Population: All participants received at least one vaccination.
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
Number analyzed (Participants) | 124 | 125 | 125
percent of participants
  SAE after any dose | 2.4 [0.5 to 6.9] | 2.4 [0.5 to 6.9] | 0.0 [0.0 to 2.9]
  Related SAE | 0.0 [0.0 to 2.9] | 0.0 [0.0 to 2.9] | 0.0 [0.0 to 2.9]

4. Primary Outcome: Percentage of Participants With AE of Special Interest by Severity and Relatedness Throughout the Entire Study Period
Description: AEs of Special interest which are AEs relevant to COVID-19 and potential immune-mediated medical conditions (PIMMC) occurred throughout the entire study period
Time Frame: From first vaccination to Day 197
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
Number analyzed (Participants) | 124 | 125 | 125
percent of participants | 0.8 [0.0 to 4.4] | 0.0 [0.0 to 2.9] | 0.0 [0.0 to 2.9]

5. Primary Outcome: NT50 GMT at 14 Days and 6 Months After Second Vaccination
Description: NT50 GMT against SARS-CoV-2 pseudovirus in subjects who are anti-S IgG seronegative at baseline
Time Frame: 14 days and 6 months after second vaccination
Population: NT50 GMTs are analyzed from subjects with seronegative anti-S IgG at baseline.
  - There were 18 subjects were sero-positive at baseline (anti-S IgG ≥50.3 ELU/mL), 2 subjects (AstraZeneca) had invalid result (IR) at Baseline (D1), 3 subjects did not received 2nd vaccination, 7 subjects were missed visit (D197), and 4 subjects had invalid result (D197)
Measure: Geometric Mean (95% Confidence Interval); unit: IU/ml
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
Number analyzed (Participants) | 120 | 118 | 114
IU/ml
  At 14 days after second vaccination | 162.78 [136.79 to 193.71] | 200.72 [166.15 to 242.47] | 93.14 [77.70 to 111.66]
  At 6 months after second vaccination: number analyzed (Participants) | 116 | 115 | 110
  At 6 months after second vaccination | 152.38 [91.74 to 253.08] | 132.48 [80.70 to 217.50] | 92.90 [60.28 to 143.18]

6. Primary Outcome: GMFR in NT50 at 14 Days and 6 Months After Second Vaccination
Description: GMFR in NT50 against SARS-CoV-2 pseudovirus measured at 14 days and 6 months after second vaccination to the baseline
Time Frame: 14 days and 6 months after second vaccination
Population: Geometric Mean Fold Rise (GMFR) is the geometric mean of the ratios of post-vaccination to the pre-first vaccination. The analysis included subjects regardless anti S IgG status at baseline.
  * Baseline (D1): 2 subjects had invalid result (IR).
  * Visit 5 (D43): 3 subject (6 μg) did not receive 2nd dose of vaccination.
  * Visit 7 (D197): 7 subjects were missed visit , 4 subjects had invalid result, 3 subject did not receive 2nd dose of vaccination
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
Number analyzed (Participants) | 124 | 123 | 122
fold rise
  At 14 days after second vaccination | 33.14 [27.82 to 39.47] | 39.93 [33.35 to 47.81] | 17.91 [14.96 to 21.43]
  At 6 months after second vaccination: number analyzed (Participants) | 120 | 119 | 116
  At 6 months after second vaccination | 30.79 [18.70 to 50.70] | 28.35 [17.67 to 47.11] | 18.69 [12.10 to 28.88]

7. Primary Outcome: Percentage of Subjects With Seroresponse in NT50 at 14 Days and 6 Months After Second Vaccination
Description: Seroresponses against SARS-CoV-2 pseudovirus as defined by a ≥ 4-fold increase from baseline
Time Frame: 14 days and 6 months after second vaccination
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
Number analyzed (Participants) | 124 | 123 | 122
percent of participants
  At 14 days after second vaccination | 91.9 [85.7 to 96.1] | 93.5 [87.6 to 97.2] | 82.0 [74.0 to 88.3]
  At 6 months after second vaccination: number analyzed (Participants) | 120 | 119 | 116
  At 6 months after second vaccination | 50.8 [41.6 to 60.1] | 47.1 [37.8 to 56.4] | 48.3 [38.9 to 57.7]

8. Secondary Outcome: IgG GMC at 14 Days and 6 Months After Second Vaccination
Description: Anti-S IgG GMC in subjects who are anti-S IgG seronegative at baseline
Time Frame: 14 days and 6 months after the second vaccination
Population: IgG GMC are analyzed from subjects with seronegative anti-S IgG at baseline.
  - There were 18 subjects were sero-positive at baseline (anti-S IgG ≥50.3 ELU/mL), 2 subjects (AstraZeneca) had invalid result (IR) at Baseline (D1), 3 subjects did not received 2nd vaccination, 7 subjects were missed visit (D197), and 4 subjects had invalid result (D197)
Measure: Geometric Mean (95% Confidence Interval); unit: BAU/ml
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
Number analyzed (Participants) | 120 | 118 | 114
BAU/ml
  At 14 days after second vaccination | 141.91 [118.54 to 169.90] | 176.19 [144.77 to 214.43] | 348.89 [294.54 to 413.27]
  At 6 months after second vaccination: number analyzed (Participants) | 118 | 117 | 110
  At 6 months after second vaccination | 129.17 [75.93 to 219.72] | 111.77 [66.33 to 188.32] | 201.52 [127.62 to 318.22]

9. Secondary Outcome: GMFR in Anti-S IgG GMC at 14 Days and 6 Months After Second Vaccination
Description: GMFR in anti-S IgG GMC measured at 14 days and 6 months after second vaccination to the baseline
Time Frame: 14 days and 6 months after the second vaccination
Population: * The analysis included subjects regardless anti S IgG status at baseline.
  * Baseline (D1): 1 subject had invalid result (IR) of anti-S IgG.
  * Visit 5 (D43): 1 subject (3 μg) had invalid result (IR) of anti-S IgG at baseline (D1), 3 subjects did not receive 2nd dose of vaccination.
  * Visit 7 (D197): 1 subject (3 μg) had invalid result (IR) of anti-S IgG at baseline (D1),7 subjects were missed visit, and 2 subjects did not receive 2nd dose of vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
Number analyzed (Participants) | 123 | 123 | 124
fold rise
  At 14 days after second vaccination | 45.13 [37.75 to 53.95] | 53.16 [43.79 to 64.52] | 100.89 [84.90 to 119.90]
  At 6 months after second vaccination: number analyzed (Participants) | 121 | 122 | 121
  At 6 months after second vaccination | 40.38 [23.92 to 68.17] | 35.82 [21.61 to 59.36] | 60.44 [38.86 to 94.00]

10. Secondary Outcome: Percentage of Subjects With Seroresponses in Anti-S IgG Concentration at 14 Days and 6 Months After Second Vaccination
Description: Seroresponses in anti-S IgG titer as defined by (1) a ≥ 4-fold increase from baseline, and (2) a ≥ 10-fold increase from baseline
Time Frame: 14 days and 6 months after the second vaccination
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
Number analyzed (Participants) | 123 | 123 | 124
percent of participants
  At 14 days after second vaccination | 99.2 [95.6 to 100] | 96.7 [91.9 to 99.1] | 99.2 [95.6 to 100]
  At 6 months after second vaccination: number analyzed (Participants) | 121 | 122 | 120
  At 6 months after second vaccination | 69.4 [60.4 to 77.5] | 77.9 [69.5 to 84.9] | 90 [83.2 to 94.7]

11. Other Pre Specified Outcome: IFN-gamma
Description: Magnitude, functionality, and Th polarization of S protein-specific T cells at 14 days and 6 months after the second vaccination relative to baseline
Time Frame: 14 days and 6 months after the second vaccination
Population: One participant missed the D197 visit
Measure: Median (95% Confidence Interval); unit: SFU/1x10^6 cells
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
Number analyzed (Participants) | 12 | 11 | 13
SFU/1x10^6 cells
  SARS-CoV-2 vial 1 - DMSO at 14 days after second vaccination | 15.00 [8.00 to 30.00] | 8.00 [3.00 to 63.00] | 60 [27.00 to 238.00]
  SARS-CoV-2 vial 1 - DMSO at 6 months after second vaccination: number analyzed (Participants) | 12 | 11 | 12
  SARS-CoV-2 vial 1 - DMSO at 6 months after second vaccination | 40.00 [10.00 to 110.00] | 30.00 [10.00 to 97.00] | 97.00 [21.00 to 180.00]
  SARS-CoV-2 vial 2 - DMSO at 14 days after second vaccination | 16.00 [3.00 to 33.00] | 11.00 [0.00 to 33.00] | 70.00 [20.00 to 187.00]
  SARS-CoV-2 vial 2 - DMSO at 6 months after second vaccination: number analyzed (Participants) | 12 | 11 | 12
  SARS-CoV-2 vial 2 - DMSO at 6 months after second vaccination | 40.00 [15.00 to 168.00] | 25.00 [20.00 to 75.00] | 60.00 [21.00 to 154.00]

12. Other Pre Specified Outcome: IL5
Description: Magnitude, functionality, and Th polarization of S protein-specific T cells relative to baseline
Time Frame: 14 days and 6 months after second vaccination
Population: One participant missed the D197 visit
Measure: Median (95% Confidence Interval); unit: SFU/1x10^6 cells
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
Number analyzed (Participants) | 12 | 11 | 13
SFU/1x10^6 cells
  SARS-CoV-2 vial 1 - DMSO at 14 days after second vaccination | 1.00 [0.00 to 2.00] | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 5.00]
  SARS-CoV-2 vial 1 - DMSO at 6 months after second vaccination | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 5.00] | 0.00 [0.00 to 2.00]
  SARS-CoV-2 vial 2 - DMSO at 14 days after second vaccination | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 3.00]
  SARS-CoV-2 vial 2 - DMSO at 6 months after second vaccination | 0.00 [0.00 to 3.00] | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 0.00]

ADVERSE EVENTS:
Time Frame: - 7 days after each vaccination for solicited AEs - 28 days after each vaccination for unsolicited AEs - From first vaccination to Day 197 for AE of special interest (AESIs) and SAE
Arm/Group | COVIVAC 3 mcg | COVIVAC 6 mcg | AZD1222
All-Cause Mortality (participants affected / at risk) | 0/124 | 0/125 | 0/125
Serious Adverse Events (participants affected / at risk) | 5/124 | 3/125 | 0/125
Other Adverse Events (participants affected / at risk) | 25/124 | 22/125 | 25/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COVIVAC 3 mcg (N=124) | COVIVAC 6 mcg (N=125) | AZD1222 (N=125)
BRAIN CONCUSSION (DUE TO TRAFFIC ACCIDENT) (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
STOMACH CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LEUKEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CHRONIC INFLAMMATION OF THE SALIVARY GLANDS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
INFECTION AFTER SURGERY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | COVIVAC 3 mcg (N=124) | COVIVAC 6 mcg (N=125) | AZD1222 (N=125)
Covid-19 (Infections and infestations) | 25 (25) | 22 (22) | 25 (25)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/94/NCT05940194/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT05940194/SAP_001.pdf